CLINICAL TRIAL: NCT07000396
Title: The Role of Mucosal Associated Invariant t Lymphocytes in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mostafa Ali, Doctor, Assiut University
Other Study IDs: MAIT Cells in Breast Cancer
Record Dates: First submitted 2025-05-24; First posted 2025-06-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: breast cancer patients
- Group B: normal individual (control)

SUMMARY:
Evaluation of MAIT cells in patient recently diagnosed as cancer breast and its correlation with clinical outcome.

Mucosal Associated Invariant T cells are a population of unconventional T cells which are enriched in mucosal tissues such as the lung and gut but are also present in other tissues including the skin, adipose tissue and the liver [4,5,6,7]. Unlike conventional T cells, MAIT cells are not restricted by MHC but recognize the MHC-related protein MR1. MAIT cells express a semi-invariant TCR α-chain (Vα7.2-Jα33/20/12 in humans) and a limited repository of TCR-β chains, mostly from the TRBV20 and TRBV6 gene families [8,9]

MAIT cells can also be activated independent of TCR engagement, via pro-inflammatory cytokines such as IL-18 [10,11,12]. Upon activation, MAIT cells can rapidly respond, producing a milieu of cytokines including interferon-gamma , tumor necrosis factor alpha and interleukin-17 [11,14]. MAIT cell cytokine profiles can vary depending on their tissue localization [15].

Peripheral MAIT cells are potent producers of IFNγ and TNFα, whereas IL-17 producing MAIT cells are rare in the periphery but are more abundant in, for example, the female genital mucosa [16]. In addition to cytokine production, A central role in immune protection against cancer is played by T lymphocytes, particularly CD8+ T cells .Their infiltration in tumor cell nests is usually associated with a favorable prognosis and may predict outcome of therapies with drugs that block immune inhibitory receptors (checkpoint blockade.

A recent meta-analysis reported that tumor-infiltrating CD8+ lymphocytes can be identified in 48% of all breast cancers .Interestingly, triple-negative breast cancers show the highest incidence of lymphocyte predominance. Moreover, TILs were found to be prognostic in triple-negative breast cancer, and higher levels of TILs were predictive for trastuzumab benefit in HER2+ disease. These findings suggest that therapies that enforce immune responses could potentially improve patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Female patients admitted at South Egypt cancer institute who diagnosed as breast cancer based on full clinical, radiologic and pathologic assays

Exclusion Criteria:

1. Patients receive any anti-cancer therapy.
2. Patients diagnosed with other concomitante cancer or chronic disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Female patients admitted at South Egypt cancer institute who diagnosed as breast cancer based on full clinical, radiologic and pathologic assays
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between mucosal associated invariant t lymphocytes and breast cancer outcome | Baseline
  The role of mucosal associated invariant t lymphocytes in breast cancer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zumwalde NA, Haag JD, Gould MN, Gumperz JE. Mucosal associated invariant T cells from human breast ducts mediate a Th17-skewed response to bacterially exposed breast carcinoma cells. Breast Cancer Res. 2018 Sep 12;20(1):111. doi: 10.1186/s13058-018-1036-5. PMID 30208917